CLINICAL TRIAL: NCT01273493
Title: An Open-Label, Multicenter, Pharmacokinetic Study of Trabectedin in Subjects With Advanced Malignancies and Hepatic Dysfunction
Brief Title: A Pharmacokinetic Study of Trabectedin in Patients With Advanced Malignancies and Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017542; ET7430OVC1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-12-23; First posted 2011-01-10 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasm Metastases; Hepatic Insufficiency
Keywords: Trabectedin, YONDELIS; Antineoplastic Agents; Solid tumors; Locally advanced or metastatic disease; Chemotherapy; Pharmacokinetics; Hepatic Dysfunction
MeSH Terms: conditions — Neoplasm Metastasis; Hepatic Insufficiency; Liver Diseases | interventions — Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trabectedin 1.3 mg/m^2 plus Dexamethasone (Experimental): Control group Trabectedin 1.3 mg/m^2 i.v.will be administered on Day 1. Dexamethasone will be administered 30 minutes prior to trabectedin.
  Interventions: Drug: Trabectedin; Drug: Dexamethasone
- Trabectedin 0.58 mg/m^2 plus Dexamethasone (Experimental): Hepatic dysfunction group Trabectedin 0.58 mg/m^2 (or adjusted dose) i.v. will be administered on Day 1. Dexamethasone will be administered 30 minutes prior to trabectedin.
  Interventions: Drug: Trabectedin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Trabectedin — Trabectedin 0.58 or 1.3 mg/m^2 (or adjusted dose) i.v. will be administered on Day 1.
Drug: Dexamethasone — Dexamethasone will be administered as 20 mg/m^2, 30 minutes prior to trabectedin.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (blood levels) of trabectedin after administration to patients with advanced malignancies and hepatic (liver) dysfunction.

DETAILED DESCRIPTION:
This is an open-label (patients will know the names of study drugs they receive), single-dose, study that will examine the pharmacokinetics (blood levels) and assess survival and safety of trabectedin in patients with advanced malignancies who either have hepatic (liver) dysfunction or do not have hepatic dysfunction (patients enrolled without hepatic dysfunction will be referred to as the control group). Trabectedin is a drug being developed to treat patients with cancer that will be administered intravenously (i.v.) through a catheter (tube) into a central vein. In addition, dexamethasone, a drug used to prevent nausea and vomiting in chemotherapy patients that may have protective effects on the liver, will be administered to patients before the administration of trabectedin. Patients who complete the treatment phase of the study who in the opinion of the investigator would derive an overall clinical benefit from further treatment with trabectedin will have the opportunity to continue treatment with trabectedin in the optional extension phase. The dose and schedule of trabectedin may be modified by the treating physician in the optional extension phase to be more appropriate for the type of malignancy being treated. A single dose of trabectedin (1.3 mg/m2 in patients in the control group and 0.58 mg/m2 in patients with hepatic dysfunction) will be administered by i.v.infusion over a 3-hour period. The dose of trabectedin may be adjusted if necessary for patients with hepatic dysfunction subsequently enrolled in the study. All patients will be administered dexamethasone 20 mg i.v. (or equivalent) approximately 30 minutes before the administration of trabectedin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic disease, any solid tumor except hepatocellular carcinoma, who have been previously treated with systemic chemotherapy (chemotherapy administered through the blood) and who have had relapsed or had progressive disease following standard of care treatment with chemotherapy prior to enrollment, or intolerant to prior standard of care treatment with chemotherapy
* Patients with Eastern Cooperative Oncology Group (ECOG) score of <=2 at the time of screening
* Patients enrolled with hepatic dysfunction must have laboratory test results for total bilirubin of >1.5x to <=3x the upper limit of normal (ULN) and liver function tests (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) of <8x the ULN
* Patients enrolled without hepatic dysfunction must have laboratory test results for total bilirubin of less than the ULN, alkaline phosphatase (ALP) <=1.5x the ULN, and AST and ALT of <=the ULN.

Exclusion Criteria:

* Patients with previous exposure to trabectedin
* Patients with known liver disease
* Patients diagnosed with hepatocellular carcinoma, or who have a history of biliary sepsis within the past 2 years
* Patients unwilling to have a central catheter
* In hepatic dysfunction group, patients with hepatic dysfunction who have Gilbert's syndrome. Patients signs of encephalopathy (altered brain function).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of trabectedin | At protocol-specified time points for up to 8 days

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to 30 days after the administration of trabectedin
Findings from clinical laboratory evaluations | Up to 30 days after the administration of trabectedin
Findings from vital signs measurements | Up to 30 days after the administration of trabectedin
Findings from physical examinations | Up to 30 days after the administration of trabectedin
Evaluate survival data | at a time point to be determined by the sponsor at a later date.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- United States (6):
  - Scottsdale, Arizona
  - Detroit, Michigan
  - New York, New York
  - Philadelphia, Pennsylvania
  - Salt Lake City, Utah
  - Tacoma, Washington
- Belgium (2):
  - Edegem
  - Wilrijk
- Edmonton, Alberta, Canada
- Spain (2):
  - Barcelona
  - Madrid

REFERENCES:
- [Derived] Calvo E, Azaro A, Rodon J, Dirix L, Huizing M, Senecal FM, LoRusso P, Yee L, Poggesi I, de Jong J, Triantos S, Park YC, Knoblauch RE, Parekh TV, Demetri GD, von Mehren M. Hepatic safety analysis of trabectedin: results of a pharmacokinetic study with trabectedin in patients with hepatic impairment and experience from a phase 3 clinical trial. Invest New Drugs. 2018 Jun;36(3):476-486. doi: 10.1007/s10637-017-0546-9. Epub 2017 Nov 27. PMID 29177975
- See also: An Open-Label, Multicenter, Pharmacokinetic Study of Trabectedin in Subjects with Advanced Malignancies and Hepatic Dysfunction — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=872&filename=CR017542_CSR.pdf